CLINICAL TRIAL: NCT01757483
Title: Effectiveness of Risk Minimisation Interventions for Ticagrelor in Canada
Brief Title: Canadian Ticagrelor Survey
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5130L00009
Record Dates: First submitted 2012-12-18; First posted 2012-12-31 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prescribers

SUMMARY:
This study is designed to evaluate the effectiveness of the current ticagrelor risk minimisation strategy in Canada through a prescriber knowledge and understanding (KAU) survey of selected important identified safety concerns (i.e., bleeding, dyspnea and drug interactions) and ASA dosage.

DETAILED DESCRIPTION:
Effectiveness of risk minimisation interventions for ticagrelor in Canada

ELIGIBILITY:
Inclusion Criteria:

- N/A (All prescribers will be contacted for participation)

Exclusion Criteria:

- Participation in a previous wave of the survey.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All physicians who have prescribed at least one dose of ticargrelor and complete the Knowledge and understanding survey
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
KAU Questionnaire: Knowledge of the 4 key safety issues pertaining to ticagrelor (adequate or inadequate for each safety issue) | 2 months

SECONDARY OUTCOMES:
KAU Questionnaire: Practice characteristics | 2 months
KAU Questionnaire: The difference in knowledge of understanding across the key safety concerns | 2 months
KAU Questionnaire: Association between prescribers' characteristics and knowledge and understanding of the key safety concerns. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yola Moride, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Research Site, Montreal, Quebec, Canada

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=483&filename=KAU_Survey_Synopsis.pdf